CLINICAL TRIAL: NCT03953027
Title: Understanding the Impact of Drug Shortages on Oncology Care Delivery
Status: Withdrawn | Type: Observational
Why Stopped: Study is not human subjects research.
Sponsor: University of Rochester NCORP Research Base (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Elaine Hill, Assistant Professor, University of Rochester
Organization: University of Rochester (Other)
Other Study IDs: URCC18004CD; NCI-2018-03601 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); URCC18004CD (Other: University of Rochester NCORP Research Base); URCC-18004CD (Other: DCP); URCC-18004CD (Other: CTEP); UG1CA189961 (NIH)
Record Dates: First submitted 2019-05-15; First posted 2019-05-16 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-04

CONDITIONS: Community Practice; Staff

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Health Services Research (surveys about drug shortages): At baseline, practice sites complete a Baseline Drug Shortage Survey and Pharmacy Baseline Survey; Drug Shortage Incident Reports are completed in real time as cancer care delivery problems occur; and the Quarterly Follow-Up Survey Number Treated Report every 3 months for one year (4 total).
  Interventions: Other: Survey Administration

INTERVENTIONS:
Other: Survey Administration — Ancillary studies

SUMMARY:
This trial studies the impact of drug shortages on oncology care delivery. Gathering information about cancer drug shortages over time may help researchers improve access to drugs during times of shortages.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To prospectively estimate the proportion of National Cancer Institute (NCI) Community Oncology Research Program (NCORP) community practices that experience a cancer care delivery problem attributable to a drug shortage of infusional therapeutic oncology drugs.

SECONDARY OBJECTIVES:

I. To prospectively estimate the rate of cancer care delivery problems attributable to a drug shortage of infusional therapeutic oncology drugs for patient populations treated with: a) all cancer drugs, b) all cancer drugs in shortage, and c) each individual cancer drug in shortage.

II. To assess strategies practices used during drug shortages (e.g., manage costs, stockpile, hire staff).

TERTIARY OBJECTIVES:

I. To assess practice factors (e.g., case mix, size, practice type) associated with the likelihood that a practice reports cancer care delivery problems.

II. To describe how practice-level strategies in response to drug shortages vary by practice characteristics.

III. To describe the possible effects on clinical trials (e.g., unable to enroll a patient or changing to an alternative treatment).

IV. To characterize cancer care delivery problems attributable to a shortage of supportive care agents.

V. To characterize cancer care delivery problems attributable to a shortage of oral anti-cancer agents.

OUTLINE: Practice sites complete a Baseline Drug Shortage Survey, Drug Shortage Incident Reports in real time as cancer care delivery problems occur, and the Quarterly Follow-Up Survey every 3 months for one year (4 total).

ELIGIBILITY:
Inclusion Criteria:

* Be a primary affiliate or sub-affiliate of an NCORP community site or minority underserved (M/U) community site that is affiliated with the University of Rochester Cancer Center (URCC) NCORP Research Base

  * Practice sites must have a valid Cancer Therapy Evaluation Program (CTEP) identification number
  * Practice sites may or may not share a pharmacy
* Provide infusional chemotherapy treatment (either inpatient or outpatient)

Exclusion Criteria:

* Practices sites without valid CTEP identification (ID)
* Practice sites that do not provide infusional chemotherapy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Be a primary affiliate or sub-affiliate of an NCORP community site or minority underserved (M/U) community site that is affiliated with the University of Rochester Cancer Center (URCC) NCORP Research Base
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-18 (Estimated)

PRIMARY OUTCOMES:
Proportion of NCORP community practices that experience a cancer care delivery problem attributable to a drug shortage of infusional therapeutic oncology drugs | Baseline up to 12 months
  Each incident is defined by the drug in shortage and by each cancer care delivery decision (e.g., whenever a recommended treatment plan is developed). All incidents are collected de-identified and aggregated to the practice site. For each drug in shortage during the year (4 quarters) of observation, will determine the number of practices reporting a care delivery problem due to each drug during any quarter and total number of practices treating patients with the drug during any quarter. Will calculate the proportion of affected practices among practices treating patients with the drug as the ratio of these two numbers. Will calculate mean, median, range and evaluate the shape of the distribution of drug specific estimates.
Change to less effective treatment | Up to 12 months
  Assessed with the Drug Shortage Incident Report. When the primary oncology team is developing a recommended treatment plan and the preferred drug is in shortage, even if the patient never was treated with the drug in shortage, this is considered a "change" for this study. The determination of "less effective" will be made by the primary oncology team. "Less effective" treatments can include those that are not the best options per guidelines through the National Comprehensive Cancer Network, the American Society of Clinical Oncology, and other organizations that establish guidelines for oncology care. Given that the primary oncology team is in charge of the patient's care, they will determine if they think the "change" is "less effective" based on their understanding of the patient's diagnosis and clinical situation.
Change to more toxic treatment | Up to 12 months
  Assessed with the Drug Shortage Incident Report. When the primary oncology team is developing a recommended treatment plan and the preferred drug is in shortage, even if the patient never was treated with the drug in shortage, this is considered a "change" for this study. The practice site staff will verify with the primary oncology team that they perceive this cancer care delivery issue (e.g., change to another drug) to be more toxic than what was intended. Whether the "change" led to a more toxic treatment or regimen will be determined by the primary oncology team. Teams can utilize their pharmacy staff to help determine if the new treatment or regimen has data to support that it would lead to higher toxicity.
Delay in treatment | Up to 12 months
  Assessed with the Drug Shortage Incident Report. Each incident is defined by the drug in shortage and by each cancer care delivery decision (e.g., whenever a recommended treatment plan is developed). Any time there is a change to a treatment regimen due to a drug shortage, the primary oncology team should determine whether or not they perceive this change to be a problem for a patient. When there is a drug shortage that results in a potential issue (e.g., missed dose), the practice site staff will verify with the primary oncology team that they actually perceived this cancer care delivery issue as a problem. The same patient may experience multiple cancer care delivery problems over the course of their treatment. Each of these problems should be reported, de-identified, as separate incidents as they occur.
Medication error/near miss | Up to 12 months
  Assessed with the Drug Shortage Incident Report. When there is a shortage of oncology drugs and there is a change in dose, administration, or drug, there can be medication errors in dose or concentration (e.g., drug was supposed to be diluted, but is not). A near miss is when the primary oncology team identifies a potential medication error but the drug was not administered to the patient. Oncology teams should rely on pharmacy staff to help identify and define medication errors and near misses.

SECONDARY OUTCOMES:
Rate of cancer care delivery problems (CCDPs) | Up to 12 months
  For each quarter and every practice, using the Quarterly Follow-Up Survey, will evaluate the rate of CCDPs as the total number of the reported CCDP incidents (numerator) per number of patients treated (denominator). To estimate the numerator, will sum numbers of reported incidents across all drugs in shortage documented in the Infusional Chemotherapy Incident Report. The total number of patients treated within the practice in the quarter (Quarterly Follow-Up Survey) will represent the denominator. To calculate the overall average estimate of the rate (dependent variable) and its 95% confidence interval, will use a generalized linear mixed model (GLMM) with a Poisson link and independent random effects random effects for sub-affiliates considered within the nested structure of National Cancer Institute (NCI) Community Oncology Research Program (NCORP) members, their affiliates and sub-affiliates.
Strategies practices use | Baseline up to 12 months
  Strategies practices use in response to drug shortages are collected in the Baseline Drug Shortage Survey and the Quarterly Follow-Up Survey. Will calculate the proportion of practices using a particular practice-level response strategy to drug shortages. This proportion will be calculated for each of the following response strategies: stockpiling, increasing staff time, purchasing from secondary markets, changing route of administration (e.g., oral), and sending patients to another institution.

OTHER OUTCOMES:
Practice factors | Baseline up to 12 months
  Defined as case mix, size, and practice type, associated with the likelihood that a practice reports cancer care delivery problems. Will use information from the Quarterly Follow-Up Survey to identify practice-level responses. For example, will identify the number of practices that stockpile drugs and divide this number by the total number of participating practices to get the estimate and 95% confidence interval (CI) of proportion of sites stockpiling. Utilizing the baseline survey, will estimate the sites' retrospective perception about the influence of drug shortages on daily cancer care delivery by asking a series of targeted questions (e.g.; extra resources, change in treatment plan, patient sent to another institution for treatment). Since the answers to questions range on Likert scale from 1-never encounter, to 5=always, for each of the questions will estimate the distribution of provided answers.
Variation in practice characteristics | Baseline up to
  Defined as how practice-level strategies in response to drug shortages vary by practice characteristics. Data will be collected. Will use data on case mix and other practice characteristics (e.g., number of physicians, practice size, practice type, racial make-up of patients, safety-net status, region) from our Registration Form, Drug Shortage Baseline Survey and Pharmacy Baseline Survey. Will use a logistic regression model to estimate the association of practice characteristics with the outcome. Additionally, to assess the effects of practice characteristics on the rate of drug shortages, the practice characteristics will be added as fixed effects to the GLMM.
Effects of drug shortages on clinical trials | Up to 12 months
  The Quarterly Follow-Up Survey asks questions about which clinical trials were affected and whether the patient was unable to enroll or was given a different treatment. Data will be collected. Using the individual Drug Shortage Incident Report will estimate how drug shortages affect clinical trials. Will estimate the proportion of practices that experience a disruption to ongoing clinical trials using methodology.
Cancer care delivery problems associated with supportive care agents | Up to 12 months
  There is a separate incident report form that will collect problems related to supportive care agents. CCDPs will be determined by the primary oncology team. Will use descriptive statistics to evaluate patterns of cancer care delivery problems associated with shortages of supportive care agents.
Cancer care delivery problems associated with oral anticancer agents | Up to 12 months
  There is a separate incident report that will collect problems related to oral anticancer agents. CCDPs will be determined by the primary oncology team. Will use descriptive statistics to evaluate patterns of cancer care delivery problems associated with shortages of oral anti cancer agents.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Hill, PhD, Principal Investigator — University of Rochester NCORP Research Base
Locations (6):
- United States (6):
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Southeast Clinical Oncology Research Program, Winston-Salem, North Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina